CLINICAL TRIAL: NCT06564090
Title: Effect on Gait Pattern During Robot Assisted Gait Training (RAGT) of End-effector Type in Burn Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HangangSHH-20
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Burns; Gait Training; Rehabilitation
Keywords: burns; gait pattern; robot assisted gait training
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome measurements, and data analysis were performed by trained and blinded outcome assessor who was not involved in the intervention. The outcome measures were evaluated before training and immediately after 8 weeks of training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- robot assisted gait training (Experimental): Morning Walk® is a new end-effector type robot developed by Hyundai Heavy Industries and Taeha Mechatronics for lower limb rehabilitation in the patients with gait disturbance.The RAGT group received RAGT with robot training for 30 minutes and conventional physiotherapy for 30 minutes per session
  Interventions: Other: robot assisted gait training; Other: conventional gait training
- conventioanl gait training (Active Comparator): The control group received conventional physiotherapy for 60 minutes per session. Conventional physiotherapy consisted of 30 minutes of therapist-assisted gait and balance training and 30 minutes of strengthening exercises. The both group patients received five training sessions per week for 8 weeks (a total of 40 sessions).
  Interventions: Other: conventional gait training

INTERVENTIONS:
Other: robot assisted gait training — Morning Walk® is a new end-effector type robot developed by Hyundai Heavy Industries and Taeha Mechatronics for lower limb rehabilitation in the patients with gait disturbance.The RAGT group received RAGT with robot training for 30 minutes and conventional physiotherapy for 30 minutes per session.
  Arms: robot assisted gait training
Other: conventional gait training — The control group received conventional physiotherapy for 60 minutes per session. Conventional physiotherapy consisted of 30 minutes of therapist-assisted gait and balance training and 30 minutes of strengthening exercises. The both group patients received five training sessions per week for 8 weeks (a total of 40 sessions).

SUMMARY:
This study aimed to investigate gait pattern and muscles power improvement of patient with gait disturbance caused by burns after end-effector type robot (Morning Walk®)-assited gait training (RAGT). This study randomly assigned 36 patients to one of two group : 30 minutes of Morning Walk® training with 30 minutes conventional physiotherapy (RAGT group) or 60 minutes of conventional physiotherapy (CON group). Five training sessions per week were given for 8 weeks. The primary outcomes were gait performance and muscles powers, which were assessed by the functional ambulation category (FAC) and the manual muscles test (MMT), respectively. The secondary outcomes included 6-minute walking test (6MWT), gait kinematic and spatiotemporal gait parameters. The results of this study is anticipated that the patients with gait disturbance receiving the RAGT might improve greater in gait performance and normal gait patterns that those trained with conventional physiotherapy.

DETAILED DESCRIPTION:
Patients with burn injuries to the lower extremities experience gait dysfunctions due to pain or joint contractures, and gait asymmetry occurs due to complications on the affected side. The persisting gait asymmetry placed these patients at risk for potential negative consequences, such as loss of bone mineral density of the affected side, overuse injury on the unaffected side due to compensatory actions, compromised postural control, and gait inefficiencies. Early gait training through physical therapy is a pivotal strategy for enhancing patients' quality of life, functional outcomes and mitigating burn-related complications. The conventional physical therapy is instrumental in fostering an increased range of motion (ROM) and mitigating contractures following burns or skin grafts. Physical therapy centers on patients' positioning, ROM, muscles strength, endurance, balance, coordination, and respiratory rehabilitation.Previous studies using end-effector type RAGT for patients with gait disturbances have demonstrated that RAGT combined with conventional physiotherapy could significantly improved walking speed, gait performance, and motor power . This study aimed to investigate gait pattern and muscles power improvement of patient with gait disturbance caused by burns after end-effector type robot (Morning Walk®)-assited gait training (RAGT).

This study randomly assigned 36 patients to one of two group : 30 minutes of Morning Walk® training with 30 minutes conventional physiotherapy (RAGT group) or 60 minutes of conventional physiotherapy (CON group). Five training sessions per week were given for 8 weeks. The primary outcomes were gait performance and muscles powers, which were assessed by the functional ambulation category (FAC) and the manual muscles test (MMT), respectively. The secondary outcomes included 6-minute walking test (6MWT), gait kinematic and spatiotemporal gait parameters. The results of this study is anticipated that the patients with gait disturbance receiving the RAGT might improve greater in gait performance and normal gait patterns that those trained with conventional physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent split thickness skin graft (STSG) at Hangang Sacred Heart Hospital
* with full or virtually full thickness involvement ( >50% of the body surface area of the lower extremity)
* aged >18 years
* with ≤ 1 functional ambulation category (FAC) score of ≤3 were included in this study.

Exclusion Criteria:

* who had fourth-degree burns (involving muscles, tendons, and bone injuries)
* severe communication disorders due to intellectual impairment and psychologic problems
* body weight > 135kg or height >195cm
* physical status that could limit physical therapy (severe deformity or contracture of limbs, open wounds, or pressure ulcers, severe osteoporosis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
functional ambulatory category | 8 weeks
  Ambulatory ability was rated by using the functional ambulatory category (FAC) scale.

SECONDARY OUTCOMES:
6 minute walking test | 8 weeks
  6MWT was performed in accordance with the standardised guidelines, and the walking course was 20 m. Patients were instructed to walk as far as possible in 6 min
gait parameters(cadence) | 8 weeks
  steps/minutes
gait parameters(gait speed) | 8 weeks
  Measure walking speed
gait parameters(step length) | 12 weeks
  Measure the distance between steps

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang sacred heart hodpital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ebid AA, Attalla AF, Ibrahim AR, Mohamdy HM. Effect of anti-gravity treadmill (Alter G) training on gait characteristics and postural stability in adult with healed burns: A single blinded randomized controlled trial. Burns. 2024 Feb;50(1):106-114. doi: 10.1016/j.burns.2023.09.004. Epub 2023 Sep 20. PMID 37798213